CLINICAL TRIAL: NCT03556397
Title: Sentinel Lymph Node Biopsy in Patients With Breast Cancer After Neoadjuvant Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: Silesian Hospital in Opava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHIR-01-sentinel; 11360/6199/1610/021554 (Other Grant/Funding Number: Ostrava University)
Record Dates: First submitted 2018-05-24; First posted 2018-06-14 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant therapy; sentinel lymph node biopsy; axillary dissection
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: The patients will be divided into four groups, according to the stage of the disease prior to neoadjuvant therapy.
Masking Description: No roles in the study will be marked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cN0 before and after neoadjuvant th., SLNB - negative, no AD (Experimental): Patients with cN0 before and after neoadjuvant therapy, SLNB - negative, without AD
  Interventions: Procedure: Sentinel lymph node biopsy (SLNB)
- cN0 before and after neoadjuvant th., SLNB - posit., AD (Experimental): Patients with cN0 before and after neoadjuvant therapy, SLNB - positive, AD (separated histological examination of lymph nodes in levels I and II)
  Interventions: Procedure: Sentinel lymph node biopsy (SLNB); Procedure: Axillary dissection
- cN1 before neoadj. th., cN0 after neoadj. th., SLNB, AD (Experimental): Patients with cN1 before neoadjuvant th., cN0 after neoadjuvant therapy, SLNB, AD (separated histological examination of lymph nodes in levels I and II)
  Interventions: Procedure: Sentinel lymph node biopsy (SLNB); Procedure: Axillary dissection
- cN1 after neoadjuvant therapy, SLNB, AD (Experimental): Patients with cN1 after neoadjuvant therapy, SLNB, AD.
  Interventions: Procedure: Sentinel lymph node biopsy (SLNB); Procedure: Axillary dissection

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy (SLNB) — Sentinel lymph node biopsy will be performed in the patients
Procedure: Axillary dissection — Axillary dissection procedure will be performed in the patients
  Arms: cN0 before and after neoadjuvant th., SLNB - posit., AD; cN1 after neoadjuvant therapy, SLNB, AD; cN1 before neoadj. th., cN0 after neoadj. th., SLNB, AD

SUMMARY:
The aim of this study is to create clear indications for Sentinel Lymph Node Biopsy (SLNB) or Axillary Dissection (AD) in women with breast carcinoma after neoadjuvant therapy by studying the false negative rate of SLNB.

DETAILED DESCRIPTION:
The main object of the study is to evaluate, whether sentinel lymph node biopsy (SLNB) at women with breast cancer after neoadjuvant therapy is a method with a high false-negative rate. Patients will be classified into groups according to histological findings during SLNB, clinical and ultrasonography (USG) findings in the axilla. The aim of this study is to create clear indications for SLNB or axillary dissection (AD). In case of extension of SLNB indications, there will be a decrease in morbidity after surgical therapy when compared to AD, which will mean a profit for the patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast carcinoma confirmed by biopsy
* neoadjuvant therapy
* examination of axillary lymph nodes clinically and by ultrasound
* surgical therapy after neoadjuvant therapy

Exclusion Criteria:

* inflammatory breast carcinoma
* incomplete neoadjuvant therapy
* previous sentinel lymph node biopsy performed on the same side of the body
* disagreement with participation in the study
* other malignities influencing the treatment of breast carcinoma
* distant metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women with a history of breast carcinoma will be enrolled in the study.
Enrollment: 61 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Clear indications for SLNB or axillary dissection | 24 months
  Clear indications for SLNB or axillary dissection (AD) in women with breast carcinoma after neoadjuvant therapy using false-negativity rate of SLNB. False-negativity rate of SLNB under 10% is acceptable for avoiding AD.

SECONDARY OUTCOMES:
Morbidity | 24 months
  Morbidity after SLNB and AD will be assessed by check-ups provided by clinicians. The result will be the percentage of patients which suffer from some complications after SLNB or AD. Common morbidity rate after AD is 20%, after SLNB 1-2%.
Changes in the Quality of Life | 24 months
  Changes in the Quality of Life will be assessed using the standardised World Health Organisation Quality of Life (WHOQOL) questionnaire.
Overall Survival | 24 months
  The overall survival (in months, years) of the patients will be assessed.
Disease-free Survival | 24 months
  The disease-free survival (in months, years) of the patients will be assessed.
Progression-free Survival | 24 months
  The progression-free survival (in months, years) of the patients will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Žatecký, MD, Principal Investigator — Silesian Hospital in Opava
Locations (2):
- Czechia (2):
  - Silesian Hospital in Opava, Opava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava-Poruba, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided to make individual participant data available to other researchers.

REFERENCES:
- [Background] Kuehn T, Bauerfeind I, Fehm T, Fleige B, Hausschild M, Helms G, Lebeau A, Liedtke C, von Minckwitz G, Nekljudova V, Schmatloch S, Schrenk P, Staebler A, Untch M. Sentinel-lymph-node biopsy in patients with breast cancer before and after neoadjuvant chemotherapy (SENTINA): a prospective, multicentre cohort study. Lancet Oncol. 2013 Jun;14(7):609-18. doi: 10.1016/S1470-2045(13)70166-9. Epub 2013 May 15. PMID 23683750
- [Background] Caudle AS, Hunt KK, Tucker SL, Hoffman K, Gainer SM, Lucci A, Kuerer HM, Meric-Bernstam F, Shah R, Babiera GV, Sahin AA, Mittendorf EA. American College of Surgeons Oncology Group (ACOSOG) Z0011: impact on surgeon practice patterns. Ann Surg Oncol. 2012 Oct;19(10):3144-51. doi: 10.1245/s10434-012-2531-z. Epub 2012 Jul 31. PMID 22847123